CLINICAL TRIAL: NCT05605691
Title: A Post-Market Study In Greece Of A Minimally Invasive Lower Eyelid Treatment Utilizing The Renuvion System
Brief Title: Post-Market Lower Eyelid Treatment With Renuvion in Greece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-22-04
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Skin Laxity
Keywords: Periorbital
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Renuvion APR System Treatment (Experimental): Subject will be treated with the Renuvion APR system in the lower eyelid (periorbital) area.
  Interventions: Device: Renuvion APR System

INTERVENTIONS:
Device: Renuvion APR System — The Renuvion Generator (K192867) is indicated for delivery of radiofrequency energy and/or helium plasma to cut, coagulate and ablate soft tissue during open and laparoscopic surgical procedures. The Renuvion APR Handpiece (K191542) is intended to be used with compatible electrosurgical generators for the delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue during open surgical procedures.
  Together, the Renuvion Generator and Handpiece are referred to as the Renuvion APR System.

SUMMARY:
This is a prospective, multi-center, non-randomized, single-arm study of up to 15 subjects treated with the Renuvion APR System. Subjects will receive treatment with the Renuvion APR System in the lower periorbital area on both sides of the face.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, single-arm study of up to 15 subjects treated with the Renuvion APR System. Subjects will receive treatment with the Renuvion APR System in the lower periorbital area on both sides of the face.

At baseline, images will be taken utilizing the site's camera system. Baseline images will be used as comparator images for follow-up images for Independent Photographic Reviewer evaluation and subject/investigator assessments.

The treatment area will be tumesced with 20 - 25ml of fluid on each side of the periorbital area.

The treatment of the periorbital area will be accessed from an incision placed in the crease of the lower lid. Two incisions will be placed in both the medial and lateral crease of the lower lid. Treatment will be performed through one incision and the second incision will be used to allow for adequate venting of helium gas. Care will be taken to undermine the tissue and to ensure the incisions communicate with each other to allow adequate venting. An optional third lower lid incision may be made as needed. The treatment plane will be above the orbicularis muscle. The treatment settings will be 20% Power, 1 LPM, and 3 Passes. Procedure data and adverse events will be captured.

Follow-up will occur 1 day, 3 days, 7 days, 30 days, 90 days, and 180 days post-procedure; images will be taken at all visits. Investigator/subjects assessments will be completed at D30, D90, and D180 visits. Subjects may also be seen back for follow-up at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, ages 18 - 75 years old.
* ASA Physical Status Classification System Class I and Class II subjects.
* Complaint of skin laxity or lines in the lower eyelid area.
* Understands and accepts the obligation not to undergo any other procedures or treatments in the areas to be treated during study participation.
* Absence of physical conditions unacceptable to the investigator.
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
* Willing and able to comply with protocol requirements, including study-required images/photos, assessments/measurements, and returning for follow-up visits.
* Willing to release rights for the use of study photos, including in publication.
* Able to read, understand, sign, and date the informed consent.
* Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.

Exclusion Criteria:

* Subjects presenting with ASA Physical Status Classification System Classes III or higher.
* Festoons in the periorbital area.
* Prior cosmetic/aesthetic fillers (hyaluronic acid, poly-l-lactic acid, calcium hydroxylapatite, et.) in the study treatment area within the past 12 months.
* Pregnant, lactating, or plans to become pregnant during study participation.
* Known hypersensitivity or allergy to tumescent anesthetic (lidocaine/ epinephrine).
* Known hypersensitivity or allergy to ibuprofen or other NSAIDS.
* Previous surgery in the study treatment area.
* Active systemic or local skin disease that may alter wound healing.
* Significant or uncontrolled medical condition that in the opinion of the investigator participation in the study may compromise the patient's health.
* History of autoimmune disease (excluding Hashimoto's thyroiditis).
* Known susceptibility to keloid formation or hypertrophic scarring.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Possesses a surgically implanted electronic device (i.e., pacemaker).
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Participation in any other investigational study within 30 days prior to consent and throughout study participation.
* Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aris Sterodimas, MD, Principal Investigator — Metropolitan General Hospital
Locations (1):
- Metropolitan General Hospital, Athens, Greece

RESULTS

PARTICIPANT FLOW:
Groups:
- Renuvion APR System Treatment: Subject will be treated with the Renuvion APR system in the lower eyelid (periorbital) area.
  Renuvion APR System: The Renuvion Generator (K192867) is indicated for delivery of radiofrequency energy and/or helium plasma to cut, coagulate and ablate soft tissue during open and laparoscopic surgical procedures. The Renuvion APR Handpiece (K191542) is intended to be used with compatible electrosurgical generators for the delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue during open surgical procedures.
  Together, the Renuvion Generator and Handpiece are referred to as the Renuvion APR System.
Period: Overall Study
Arm/Group | Renuvion APR System Treatment
Started | 16
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Greece | 16
NRS for Pain [Count of Participants; unit: Participants]
  0 | 16
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0
Snap-Back Test Grade [Count of Participants; unit: Participants] — This test provides relative lower lid laxity. In normal lids, the skin snaps-back to the original position immediately; the longer it takes, the more laxity is present. Grade 0 (Normal lid that returns to position immediately on release), Grade I (Approx 2-3 seconds to return to original position), Grade II (4-5 seconds to return to original position), Grade III (>5 seconds but does return to original position with blinking), Grade IV (never returns to original position and continues to hand down in frank ectropion after the snap-back test).
  Participants
    Grade 0 | 0
    Grade I | 9
    Grade II | 3
    Grade III | 4
    Grade IV | 0
Medial Canthal Laxity Test Grade [Count of Participants; unit: Participants] — This test provides medial canthal laxity by means of measuring displacement. The greater the distance, the more the laxity. To perform the medial canthal laxity test, pull the lower lid laterally away from the medial canthus and measure displacement of medial punctum. Grade 0 (<2mm displacement), Grade I (approx 2mm displacement), Grade II (approx 3mm displacement), Grade III (>3mm displacement), Grade IV (does not return to baseline after release and blinking).
  Participants
    Grade 0 | 1
    Grade I | 14
    Grade II | 1
    Grade III | 0
    Grace IV | 0
Lateral Canthal Laxity Test Grade [Count of Participants; unit: Participants] — This test provides lateral canthal laxity by means of measuring displacement. The greater the distance, the more the laxity. To perform the lateral canthal laxity test, pull the lower lid medially away from the lateral canthus and measure displacement of lateral canthal corner. Grade 0 (<2mm displacement), Grade I (2-4mm displacement), Grade II (4-6mm displacement), Grade III (>6mm displacement), Grade IV (does not return to baseline after release and blinking).
  Participants
    Grade 0 | 1
    Grade I | 14
    Grade II | 1
    Grade III | 0
    Grade IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Day 180 Number of Participants With Improvement in Lower Eyelid Area as Determined by a Masked, Qualitative Assessment.
Description: Improvement in the lower eyelid area as determined by a masked, qualitative assessment of photographs at 180-days post-treatment compared to baseline by blinded independent reviewers. Improvement will be assessed based on photographs taken at all visits using the site's 2D camera system.
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants | 5

2. Secondary Outcome: Day 90 Number of Participants With Improvement in the Lower Eyelid Area as Determined by a Masked, Qualitative Assessment.
Description: Improvement in the lower eyelid area as determined by a masked, qualitative assessment of photographs at 90-days post-treatment compared to baseline by blinded independent reviewers. Improvement will be assessed based on photographs taken at all visits using the site's 2D camera system.
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants | 8

3. Other Pre Specified Outcome: Snap-Back Test Grade Analysis of Change From Baseline to Day 30
Description: This test provides relative lower lid laxity. In normal lids, the skin snaps-back to the original position immediately; the longer it takes, the more laxity is present. To perform the snap-back test, pull the lower lid away and down from globe for several seconds and wait to see how long it returns to the original position without the subject blinking. Grade 0 (Normal lid that returns to position immediately on release), Grade I (Approx 2-3 seconds to return to original position), Grade II (4-5 seconds to return to original position), Grade III (>5 seconds but does return to original position with blinking), Grade IV (never returns to original position and continues to hand down in frank ectropion after the snap-back test).
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

4. Other Pre Specified Outcome: Snap-Back Test Grade Analysis of Change From Baseline to Day 90
Description: as for outcome 3
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

5. Other Pre Specified Outcome: Snap-Back Test Grade Analysis of Change From Baseline to Day 180
Description: as for outcome 3
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

6. Other Pre Specified Outcome: Medical Canthal Laxity Test Analysis of Change From Baseline to Day 30
Description: This test provides medial canthal laxity by means of measuring displacement. The greater the distance, the more the laxity. To perform the medial canthal laxity test, pull the lower lid laterally away from the medial canthus and measure displacement of medial punctum. Grade 0 (<2mm displacement), Grade I (approx 2mm displacement), Grade II (approx 3mm displacement), Grade III (>3mm displacement), Grade IV (does not return to baseline after release and blinking).
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 13
  Grade I | 2
  Grade II | 0
  Grade III | 0
  Grade IV | 0

7. Other Pre Specified Outcome: Medical Canthal Laxity Test Analysis of Change From Baseline to Day 90
Description: as for outcome 6
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

8. Other Pre Specified Outcome: Medical Canthal Laxity Test Analysis of Change From Baseline to Day 180
Description: as for outcome 6
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

9. Other Pre Specified Outcome: Lateral Canthal Laxity Test Analysis of Change From Baseline to Day 30
Description: This test provides lateral canthal laxity by means of measuring displacement. The greater the distance, the more the laxity. To perform the lateral canthal laxity test, pull the lower lid medially away from the lateral canthus and measure displacement of lateral canthal corner. Grade 0 (<2mm displacement), Grade I (2-4mm displacement), Grade II (4-6mm displacement), Grade III (>6mm displacement), Grade IV (does not return to baseline after release and blinking).
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 13
  Grade I | 2
  Grade II | 0
  Grade III | 0
  Grade IV | 0

10. Other Pre Specified Outcome: Lateral Canthal Laxity Test Analysis of Change From Baseline to Day 90
Description: as for outcome 9
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

11. Other Pre Specified Outcome: Lateral Canthal Laxity Test Analysis of Change From Baseline to Day 180
Description: as for outcome 9
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Grade 0 | 15
  Grade I | 0
  Grade II | 0
  Grade III | 0
  Grade IV | 0

12. Other Pre Specified Outcome: Subject Modified Global Aesthetic Improvement Scale (GAIS)
Description: The subject will grade the overall improvement of treatment area as very much improved, much improved, improved, no change, worse, much worse, and very much worse.
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 14
  Much Improved | 1
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

13. Other Pre Specified Outcome: Subject Modified Global Aesthetic Improvement Scale (GAIS)
Description: as for outcome 12
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 10
  Much Improved | 5
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

14. Other Pre Specified Outcome: Investigator Modified Global Aesthetic Improvement Scale (GAIS)
Description: The investigator will grade the overall improvement of treatment area as very much improved, much improved, improved, no change, worse, much worse, and very much worse.
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 15
  Much Improved | 0
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

15. Other Pre Specified Outcome: Investigator Modified Global Aesthetic Improvement Scale (GAIS)
Description: as for outcome 14
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 14
  Much Improved | 1
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

16. Other Pre Specified Outcome: Day 180 Patient Satisfaction Questionnaire (PSQ)
Description: At Day 180 Follow-Up visit, the study subjects will be asked to complete a subject satisfaction survey referring to the assessment of baseline photos, current photos, and a hand mirror. Yes/No - did you notice any improvement in your lower eyelid area? If yes, checkbox - improvement in wrinkles, less sagging skin, smother skin texture, other. How would you characterize your satisfaction with the treatment - very satisfied, satisfied, slightly satisfied, neither satisfied or dissatisfied, slightly dissatisfied, dissatisfied, very dissatisfied. Yes/No - would you recommend this treatment to your friends and family members.
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  Improvement Noticed: Yes | 15
  Improvement Noticed: No | 0
  Improvement in Wrinkles: Yes | 7
  Improvement in Wrinkles: No | 8
  Less Sagging Skin: Yes | 12
  Less Sagging Skin: No | 3
  Smoother Skin Texture: Yes | 11
  Smoother Skin Texture: No | 4
  Level of Satisfaction (Very Satisfied, Satisfied, Slightly Satisfied): Yes | 15
  Level of Satisfaction (Very Satisfied, Satisfied, Slightly Satisfied): No | 0
  Yes, would recommend to friends & family: Yes | 15
  Yes, would recommend to friends & family: No | 0

17. Other Pre Specified Outcome: Average Pain at Procedure Day Reported by Subject
Description: Study subjects will be asked to complete a 11-point Numeric Rating Scale (NRS) for the level of pain and discomfort associated with the study procedure. Rating Scale where 0 is "No Pain" and 10 is "Worst Possible Pain"
Time Frame: Procedure Day 0 Following Study Treatment (within 60 minutes post procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 16
Participants
  0 | 16
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

18. Other Pre Specified Outcome: Average Pain at Day 1 Reported by Subject
Description: as for outcome 17
Time Frame: 1-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 16
Participants
  0 | 16
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

19. Other Pre Specified Outcome: Average Pain at Day 3 Reported by Subject
Description: as for outcome 17
Time Frame: 3-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 16
Participants
  0 | 16
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

20. Other Pre Specified Outcome: Average Pain at Day 7 Reported by Subject
Description: as for outcome 17
Time Frame: 7-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 16
Participants
  0 | 16
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

21. Other Pre Specified Outcome: Average Pain at Day 30 Reported by Subject
Description: as for outcome 17
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

22. Other Pre Specified Outcome: Average Pain at Day 90 Reported by Subject
Description: as for outcome 17
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

23. Other Pre Specified Outcome: Average Pain at Day 180 Reported by Subject
Description: as for outcome 17
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System Treatment
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

ADVERSE EVENTS:
Time Frame: Through Day 180 follow-up visit.
Description: Adverse events and expected treatment effects (ETEs) were collected.
Arm/Group | Renuvion APR System Treatment
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renuvion APR System Treatment (N=16)
Bruise (ETE) (Skin and subcutaneous tissue disorders) | 14 (14) — Expected Treatment Effect
Contact Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Edema (ETE) (Skin and subcutaneous tissue disorders) | 13 (13) — Expected Treatment Effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05605691/Prot_SAP_000.pdf